CLINICAL TRIAL: NCT01076413
Title: Comparison of Two Exercise Interventions to Improve Gait in Older Persons: The PRIME (Program to Improve Mobility in The Elderly) Study
Brief Title: Comparison of Two Exercise Interventions to Improve Gait in Older Persons
Acronym: PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer S. Brach, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO09080228; K23AG026766 (NIH)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Gait
Keywords: gait; exercise; skill-based; aerobic
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- skill-based exercise (Experimental): 2 times per week for 12 weeks. warm-up, stretching, strengthening, and skill-based exercises. Pre-gait and gait activities including stepping patterns and walking patterns and treadmill training at various walking speeds
  Interventions: Behavioral: skill based exercise
- aerobic exercise training (Active Comparator): warm-up, strengthening and aerobic conditioning (treadmill walking)
  Interventions: Behavioral: aerobic conditioning

INTERVENTIONS:
Behavioral: skill based exercise — 2 times per week for 12 weeks Pre gait and gait activities
  Arms: skill-based exercise
Behavioral: aerobic conditioning — 2 times per week for 12 weeks. aerobic conditioning exercise consisting of treadmill walking
  Arms: aerobic exercise training

SUMMARY:
The purpose of this research study is to compare two different exercise treatments for walking problems in older adults. The investigators want to determine if participation in the exercise programs for 3 months will improve walking abilities by improving balance and strength.

DETAILED DESCRIPTION:
The purpose of this research study is to compare two different exercise treatments for walking problems in older adults. We want to determine if participation in the exercise programs for 3 months will improve walking abilities by improving balance and strength.

Adults aged 65 years or older, who are able to walk without the help of another person, are being asked to participate. If you are able to walk independently and you have medical clearance from your physician to participate in activities requiring low to moderate physical activity, you are invited to participate. We plan to enroll 40 older adults, all who have small problems with walking due to balance or strength, in this research study.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age and older
2. Ambulatory without an assistive device or the assistance of another person
3. Usual 4 meter gait speed ≥1.0 m/s
4. Completes a figure-of-eight walk in > 8.0 seconds

Exclusion Criteria:

1. Inability to participate in testing:

   1. persistent lower extremity pain that is present on most days of the week and crepitus, tenderness or enlargement of joints of the lower extremity (arthritis).84
   2. back pain that is present on most days of the weeks and interferes with walking and activities of daily living or back pain that increases with walking (lumbar stenosis)
   3. calf pain or cramping which worsens with walking and is relieved by rest (PAD)
   4. refusal to walk on a treadmill
2. Safety concerns:

   1. dyspnea at rest or during activities of daily living or use supplemental oxygen (CHF, COPD)
   2. any acute illness or medical condition that is not stable according to the approving physician
   3. resting systolic blood pressure ≥ 200 mm Hg or diastolic blood pressure ≥ 100 mm Hg or resting heart rate > 100 or < 40 beats per minute85
   4. diagnosed dementia or cognitive impairment defined as a MMSE score < 24
   5. hospitalized in the past 6 months for acute illness or surgery, other than minor surgical procedures
   6. severe visual impairment with visual acuity < 20/70 with best correction
   7. history of stroke
   8. fixed or fused lower extremity joints such as hip, knee or ankle
   9. lower extremity strength <4/5 on manual muscle testing
   10. lower extremity amputation
   11. progressive movement disorder such as MS, ALS or Parkinson's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Gait | 12 weeks
  gait characteristics, smoothness of walking, 6 MWT, complex walking tests, GARS-M, SPPB, energy cost, SAFFE, GES, figure of 8
Physical function | 12 weeks
  LLFDI function and disability scales
Physical Activity | 12 weeks
  Actigraph accelerometer

SECONDARY OUTCOMES:
Disability and health care costs | 6 months post exercise
  Late Life Function and disability index, fall history and health care cost questionnaire will be administered through a phone interview 6 months following completion of the exercise program

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Brach JS, Lowry K, Perera S, Hornyak V, Wert D, Studenski SA, VanSwearingen JM. Improving motor control in walking: a randomized clinical trial in older adults with subclinical walking difficulty. Arch Phys Med Rehabil. 2015 Mar;96(3):388-94. doi: 10.1016/j.apmr.2014.10.018. Epub 2014 Nov 10. PMID 25448244
- [Result] Brach JS, Van Swearingen JM, Perera S, Wert DM, Studenski S. Motor learning versus standard walking exercise in older adults with subclinical gait dysfunction: a randomized clinical trial. J Am Geriatr Soc. 2013 Nov;61(11):1879-86. doi: 10.1111/jgs.12506. Epub 2013 Oct 28. PMID 24219189